CLINICAL TRIAL: NCT03893591
Title: A Prospective Cohort Study to Examine the Need to Adjust the Dose of Anticoagulant Apixaban When Used in Patients With Atrial Fibrillation and Obesity
Brief Title: A Prospective Study to Examine the Need to Adjust the Dose of Apixaban When Used in Atrial Fibrillation and Obesity
Status: Completed | Type: Observational
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Lee Goldstein, Principal Investigator, HaEmek Medical Center, Israel
Other Study IDs: 0004-19
Record Dates: First submitted 2019-03-26; First posted 2019-03-28 (Actual); Last update posted 2020-04-01 (Actual); Status verified 2020-03

CONDITIONS: Anticoagulant; Apixaban; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Body mass index below 35
  Interventions: Diagnostic Test: Anti Xa levels
- Body mass index 35 and above
  Interventions: Diagnostic Test: Anti Xa levels

INTERVENTIONS:
Diagnostic Test: Anti Xa levels — one Blood sample

SUMMARY:
A prospective cohort study to determine whether a high body weight (BMI equal to or greater than 35 kg / m 2) has an effect on anticoagulant Apixaban level in the blood of patients with atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

- hospitalized Patients on Steady State level of Apixaban, based on the data given in the hospital ward . A level of Steady State is received within two days of treatment.

Exclusion Criteria:

* Anasarca
* acute renal failure

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: adults
Sampling Method: Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
Anti Xa level of patients with atrial fibrillation and obesity while treatment of Apixaban. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- HaEmek Medical Center, Afula, Israel

IPD SHARING:
Plan to Share IPD: No